CLINICAL TRIAL: NCT07367568
Title: Comparison of Costotransverse Foramen Block With Erector Spinae Plane Block in Modified Radical Mastectomy: A Randomized Controlled Trial
Brief Title: Costotransverse Foramen Block With Erector Spinae Plane Block in Modified Radical Mastectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Mai Mohamed El Rawas, Assistant professor of Anaesthesia, Intensive Care and Pain Management, National Cancer Institute, Cairo University Cairo University, Cairo, Egypt., National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP2509-501-124-203
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Costotransverse Foramen Block; Erector Spinae Plane Block; Modified Radical Mastectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTFB Group (Experimental): Patients will receive an ipsilateral ultrasound-guided costotransverse foramen block with injection of 20 ml bupivacaine 0.25%.
  Interventions: Other: Costotransverse foramen block
- ESPB Group (Experimental): Patients will receive an ipsilateral ultrasound-guided erector spinae plane block with injection of 20 ml bupivacaine 0.25%.
  Interventions: Other: Erector spinae plane block

INTERVENTIONS:
Other: Costotransverse foramen block — Patients will receive an ipsilateral ultrasound-guided costotransverse foramen block with injection of 20 ml bupivacaine 0.25%.
  Arms: CTFB Group
Other: Erector spinae plane block — Patients will receive an ipsilateral ultrasound-guided erector spinae plane block with injection of 20 ml bupivacaine 0.25%.
  Arms: ESPB Group

SUMMARY:
This study aims to compare the costotransverse foramen block with erector spinae plane block in modified radical mastectomy.

DETAILED DESCRIPTION:
Postoperative pain following modified radical mastectomy (MRM) is a considerable consequence, impacting the ipsilateral upper limbs, axillae, and thorax, resulting in diminished functional ability and substantial economic and societal repercussions.

Erector spinae plane block (ESPB), an interfascial block, minimizes nerve and vessel injury by allowing local anesthetics to diffuse across relevant spaces; it is technically simpler and has shown benefits in reducing postoperative analgesic use and pain scores.

A novel technique, the costotransverse foramen block (CTFB), is one type of Inter-transverse process (ITP) blocks. This technique entails the anterior dispersion of the local anesthetic injectate into the paravertebral region, affecting the thoracic nerve at the injection site and neighboring levels, while exhibiting negligible posterior diffusion of dye to the deep back muscles

ELIGIBILITY:
Inclusion Criteria:

* Adult females > 18 years and ≤ 65 years old.
* American Society of Anesthesiologists (ASA) physical status П-III.
* Body mass index (BMI) 18-35 kg/m2.
* Scheduled for modified radical mastectomy.

Exclusion Criteria:

* Known allergy or hypersensitivity to local anesthetic agents.
* Active infection at the injection site (e.g., cellulitis, abscess).
* Coagulopathy or ongoing anticoagulant/antiplatelet therapy [International Normalized Ratio (INR) > 1.5 or platelet count < 100,000/µL].
* Severe respiratory, cardiac, hepatic, or renal disease.
* Morbid obesity.
* Severe cognitive impairment or uncooperative behavior that could interfere with block placement.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females scheduled for modified radical mastectomy
Enrollment: 110 (Estimated)
Dates: Start 2026-01-24 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  If the numeric rating scale (NRS) is ≥ 4, an IV morphine dose (3 mg) will be provided Paracetamol 1 gm and ketorolac 30 mg will be administered every 8 hours postoperatively.

SECONDARY OUTCOMES:
Degree of pain | 48 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS) score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS score will be recorded in post-anesthesia care unit (PACU) then at 1, 6, 12, 18, 24, and 48 hours postoperatively.
Time to first request of rescue analgesia | 24 hours postoperatively
  Time to first request of rescue analgesia will be recorded from the end of surgery till first dose of morphine administrated.
Intraoperative fentanyl consumption | Intraoperatively
  Intraoperative fentanyl consumption will be recorded.
Mean arterial pressure | 4 hours postoperatively
  Mean arterial pressure will be recorded immediately before induction of anesthesia, 15 min after performing the block incision and at 20-minute intervals intraoperatively, and then hourly till 4 hours postoperatively.
Heart rate | 4 hours postoperatively
  Heart rate will be recorded immediately before induction of anesthesia, 15 min after performing the block incision and at 20-minute intervals intraoperatively, and then hourly till 4 hours postoperatively.
Incidence of adverse effects | 24 hours postoperatively
  Incidence of adverse effects such as nausea, vomiting, hypotension, and bradycardia, pneumothorax, local anesthetic toxicity for up to 24 hours post-surgery will be documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.